CLINICAL TRIAL: NCT02467101
Title: Prospective Double-blind, Placebo Controlled Study to Assess the Efficacy of Intralesional Corticoid on the Treatment of Frontal Fibrosing Alopecia
Brief Title: Study to Assess the Efficacy of Intralesional Corticosteroid on the Treatment of Frontal Fibrosing Alopecia
Acronym: FFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rubina Alves (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor-Investigator, Rubina Alves, Specialist Dermatology, M.D., Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UIC-FFA; UICatalunya (Registry Identifier: Rubina Alves)
Record Dates: First submitted 2015-05-27; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Frontal Fibrosing Alopecia
Keywords: cicatricial alopecia; treatment; placebo; double-blind
MeSH Terms: conditions — Alopecia | interventions — Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corticosteroid/Saline (Experimental): Corticosteroid/Saline
  Patients with diagnosis of frontal fibrosing alopecia are included in the study. The diagnosis is based on the clinical findings of frontal and temporoparietal hairline recession with loss of follicular ostia.
  In the same patient, intralesional triamcinolone acetone will be injected to half-head (in the active border of hairline) and in the other half-head the patient will be injected with saline solution (placebo).
  The intralesional triamcinolone acetone (40 mg/ml)l) of 0,1 mL/1cm, is given along the frontal and frontoparietal hairline every 4 weeks (3 sessions).
  This study includes 4 visits: 3 visits of treatment (with 1-month interval) and 1 visit of follow-up (month 6).
  Interventions: Other: Corticosteroid/Saline

INTERVENTIONS:
Other: Corticosteroid/Saline — Corticosteroid/Saline
  Two groups were defined: group A and group B.
  * Group A receives treatment with intralesional triamcinolone acetonide on the right half-head and placebo on the left half-head
  * Group B receives administration of intralesional triamcinolone acetonide on left half-head and placebo on the right half-head.
  Same patient will be injected with intralesional triamcinolone acetonide and a saline solution.
  Each patient will be injected on half-head.
  Other Names: Frontal fibrosing alopecia; Cicatricial alopecia; Alopecia; Hair loss

SUMMARY:
The purpose of this study is to determine the efficacy of treatment with intralesional injection of corticosteroids on the treatment of Frontal Fibrosing Alopecia (compared with placebo), between three months, six months and baseline.

DETAILED DESCRIPTION:
Frontal fibrosing alopecia (FFA) is a primary lymphocytic cicatricial alopecia, that was first described in postmenopausal women, by Kossard in 1994. Since then, FFA has also been reported in premenopausal women and rarely in men.

The exact cause of FFA is unknown. One possible reason can be the disturbed immune response to some component of the scalp hair follicles, however, whether or not the hair loss is caused by hormonal fluctuations is under question. Some authors, consider that FFA is a variant of liquen planopilaris (LPP). Whether FFA is truly an LPP variant or is a distinct entity with shared clinical features remains to be determined. FFA was also diagnosed in family members (mother and daughter) suggesting a possible genetic contribution.

Clinically, it is characterized by progressive frontal and temporoparietal recession of the hairline due to inflammatory destruction of hair follicles. Hair loss occurs in a band-like distribution and the depth of recession can be from 0,5-8 cm. Often, a small number of isolated hairs are spared within the band of alopecia.

Loss of eyebrows (partial or complete) is a finding in FFA and in some cases, can precede the hairline recession. The affected skin is atrophic, shiny, and often lighter than the chronically sun-exposed forehead skin.

The diagnosis of FFA is usually made on the basis of clinical findings, and laboratory tests are rarely required. Dermoscopy, a noninvasive tool can help for the diagnosis of FFA; The dermoscopic features of FFA are: Absence of follicular openings, perifollicular scale, and a feeble perifollicular erythema. Perifollicular erythema at the receding hairline may be a sign of active disease.

Since the first description of FFA, many reports have been published, and the number of new cases of FFA appears to be increasing.

Currently, there are no evidence-based studies to guide treatment and there is no clearly defined line of treatment for the condition. Therefore treatment options vary among clinicians.

The aim of this study is to find if intralesional triamcinolone acetonide (compared to area treated with placebo) may help to halt or slow down the progression of this disease.

The patients are divided into two groups (A and B):

1. Group A: right half-head (active border of the disease): treatment with intralesional triamcinolone acetonide left half-head (active border of the disease): placebo (saline solution)
2. Group B: right half-head (active border of the disease):placebo (saline solution)

left half-head (active border of the disease): intralesional triamcinolone acetonide

The aim of this study is to find if intralesional triamcinolone may help to halt or slow down the progres- sion of this disease.

All patients provide written informed consent before participating in the study, which is performed according to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Frontal Fibrosing Alopecia

Exclusion Criteria:

* Pregnancy
* Patient unable to accomplishing all fases of treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Phototricogram of two areas of the scalp | 6 months
  Measuring hair count (number of hairs/0.65 cm2) by comparison with 6 months and baseline

SECONDARY OUTCOMES:
Global photographs of the scalp | 6 months
  The evaluation of hair growth will be assessed by comparison of standardized images between baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Alves, M.D., Principal Investigator — Universitat Internacional Catalunya; Juan Antonio Moreno, M.D., Principal Investigator — Universitat Internacional Catalunya; Ramon Grimalt, M.D.; PhD, Study Director — Universitat Internacional Catalunya
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Barcelona, Spain